CLINICAL TRIAL: NCT00121992
Title: Phase III Randomized Comparing Docetaxel, Doxorubicin and Cyclophosphamide (TAC) vs 5-Fluorouracil, Doxorubicin and Cyclophosphamide (FAC) as Adjuvant Treatment of High Risk Operable Breast Cancer Patients With Negative Axillary Lymph Nodes
Brief Title: Docetaxel, Doxorubicin (A), Cyclophosphamide (C) (TAC) vs 5-Fluorouracil, A, C (5FAC) Breast Cancer Adjuvant Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 9805; TAX.ES1.301 (Other: RHÔNE-POULENC RORER, S.A. (RPR))
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Neoplasms
Keywords: High risk node negative breast cancer; Disease-Free survival; Quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Fluorouracil; Doxorubicin; Cyclophosphamide

ARMS (2):
- Arm A: FAC (Active Comparator): FAC (5-fluorouracil, doxorubicin, cyclophosphamide): 5-fluorouracil 500 mg/m2 iv on day 1, each 3 weeks, in combination with doxorubicin 50 mg/m2 iv and cyclophosphamide 500 mg/m2 iv
  Interventions: Drug: 5-fluorouracil; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm B: TAC (Experimental): TAC (docetaxel, doxorubicin, cyclophosphamide): Docetaxel 75 mg/m2 iv on day 1, each 3 weeks, in combination with doxorubicin 50 mg/m2 iv and cyclophosphamide 500 mg/m2 iv
  Interventions: Drug: Docetaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere
  Arms: Arm B: TAC
Drug: 5-fluorouracil
  Other Names: Adrucil
  Arms: Arm A: FAC
Drug: Doxorubicin
  Other Names: adriamycin
Drug: Cyclophosphamide
  Other Names: cytoxan

SUMMARY:
This is a prospective, non-blinded randomized phase III trial. Patients will be post-surgically stratified at inclusion first according to the participating institution, then according to menopausal status and will be randomly assigned to receive either:

* TAC: Docetaxel 75 mg/m2 as a 1 hour intravenous (i.v.) infusion on day 1 every 3 weeks (q3w) in combination with doxorubicin 50 mg/m2 as an i.v. bolus and cyclophosphamide 500 mg/m2 as an i.v. bolus on day 1 every 3 weeks.
* FAC: 5-fluorouracil 500 mg/m2 as an i.v. bolus on day 1 every 3 weeks in combination with doxorubicin 50 mg/m2 as an i.v. bolus and cyclophosphamide 500 mg/m2 as an i.v. bolus on day 1 every 3 weeks.

DETAILED DESCRIPTION:
Primary objective:

* To compare disease-free survival (DFS) after treatment with docetaxel in combination with doxorubicin and cyclophosphamide (TAC) to 5-Fluorouracil in combination with doxorubicin and cyclophosphamide (FAC) as adjuvant treatment of high risk operable breast cancer patients with negative axillary lymph nodes.

Secondary objectives:

* To compare overall survival (OS) between the 2 above mentioned arms.
* To compare toxicity and quality of life between the 2 above mentioned arms.
* To evaluate pathologic markers for predicting efficacy (hormonal receptors and human epidermal growth factor receptor 2 (HER2) protein expression).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Operable breast cancer patients (T1-T3) with negative axillary lymph nodes (10 axillary nodes dissection) and high risk criteria according to St. Gallen consensus criteria.
* Histologically proven breast cancer. Interval between surgery and registration is less than 60 days.
* Definitive surgical treatment must be either mastectomy, or breast conservative surgery. Margins of resected specimen from surgery must be histologically free of invasive adenocarcinoma and ductal carcinoma in-situ (DCIS). Lobular carcinoma in-situ is not considered as positive margin.
* Patients without proven metastatic disease.
* Estrogen and progesterone receptors performed on the primary tumour prior to randomization.
* Age between 18 years and 70 years.
* Karnofsky performance status index > 80 %.
* Adequate hepatic, renal and heart functions.
* Adequate hematology levels.
* Negative pregnancy test

Exclusion Criteria:

* Prior systemic anticancer therapy for breast cancer (immunotherapy, hormonotherapy, chemotherapy).
* Prior anthracycline therapy or taxoids (paclitaxel, docetaxel) for any malignancy.
* Prior radiation therapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant, or lactating patients.
* Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment .
* Any T4 or N1-3 or M1 breast cancer.
* Pre-existing motor or sensory neurotoxicity of a severity grade 2 by NCI criteria.
* Other serious illness or medical condition
* Past or current history of neoplasm other than breast carcinoma.
* Ipsilateral ductal carcinoma in-situ (DCIS) of the breast.
* Lobular carcinoma in-situ (LCIS) of the breast.
* Chronic treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment should be stopped before study entry.
* Definite contraindications for the use of corticosteroids.
* Concurrent treatment with other experimental drugs.
* Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.
* Male patients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 1999-07 (Actual); Primary Completion 2010-12-02 (Actual); Study Completion 2013-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario San Carlos
Locations (1):
- Spanish Breast Cancer Research Group, San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- [Background] Martin M, Pienkowski T, Mackey J, Pawlicki M, Guastalla JP, Weaver C, Tomiak E, Al-Tweigeri T, Chap L, Juhos E, Guevin R, Howell A, Fornander T, Hainsworth J, Coleman R, Vinholes J, Modiano M, Pinter T, Tang SC, Colwell B, Prady C, Provencher L, Walde D, Rodriguez-Lescure A, Hugh J, Loret C, Rupin M, Blitz S, Jacobs P, Murawsky M, Riva A, Vogel C; Breast Cancer International Research Group 001 Investigators. Adjuvant docetaxel for node-positive breast cancer. N Engl J Med. 2005 Jun 2;352(22):2302-13. doi: 10.1056/NEJMoa043681. PMID 15930421
- [Result] Martin M, Segui MA, Anton A, Ruiz A, Ramos M, Adrover E, Aranda I, Rodriguez-Lescure A, Grosse R, Calvo L, Barnadas A, Isla D, Martinez del Prado P, Ruiz Borrego M, Zaluski J, Arcusa A, Munoz M, Lopez Vega JM, Mel JR, Munarriz B, Llorca C, Jara C, Alba E, Florian J, Li J, Lopez Garcia-Asenjo JA, Saez A, Rios MJ, Almenar S, Peiro G, Lluch A; GEICAM 9805 Investigators. Adjuvant docetaxel for high-risk, node-negative breast cancer. N Engl J Med. 2010 Dec 2;363(23):2200-10. doi: 10.1056/NEJMoa0910320. PMID 21121833
- See also: home page of the Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the different subsets ("Hormone-receptor Positive and HER2 PositiveStatus Subjects", "Hormonal Receptor Positive and HER2 Negative Subjects", etc.), were assessed by central determination, and no all patients had tumor sample available.
Groups:
- Arm A: FAC: FAC (5-fluorouracil, doxorubicin, cyclophosphamide): 5-fluorouracil 500 mg/m2 iv on day 1, each 3 weeks, in combination with doxorubicin 50 mg/m2 iv and cyclophosphamide 500 mg/m2 iv
  5-fluorouracil
  Doxorubicin
  Cyclophosphamide
- Arm B: TAC: TAC (docetaxel, doxorubicin, cyclophosphamide): Docetaxel 75 mg/m2 iv on day 1, each 3 weeks, in combination with doxorubicin 50 mg/m2 iv and cyclophosphamide 500 mg/m2 iv
  Docetaxel
  Doxorubicin
  Cyclophosphamide
Period: Overall Study
Arm/Group | Arm A: FAC | Arm B: TAC
Started | 521 | 539
Hormone-receptor Positive and HER2 Positive Status Subjects | 28 | 30
Hormone-receptor Negative and HER2 Positive Status Subjects | 24 | 22
Hormone-receptor Positive and HER2 Negative Status Subjects | 209 | 220
Hormone-receptor Negative and HER2 Negative Status Subjects | 92 | 103
Completed | 519 | 528
Not Completed | 2 | 11
Not completed — Treatment not received | 2 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: FAC | Arm B: TAC | Total
Number analyzed (Participants) | 521 | 539 | 1060
Age, Continuous [Median (Full Range); unit: years] | 49 [23 to 73] | 50 [23 to 74] | 49 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521 | 539 | 1060
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 475 | 487 | 962
  Germany | 26 | 30 | 56
  Poland | 20 | 22 | 42
Tumor size [Count of Participants; unit: Participants]
  ≤2 cm | 249 | 285 | 534
  >2 to 5 cm | 258 | 241 | 499
  >5 cm | 13 | 13 | 26
  Unknown | 1 | 0 | 1
Tumor grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    Grade 1 | 34 | 38 | 72
    Grade 2 | 230 | 216 | 446
    Grade 3 | 231 | 259 | 490
    Unknown | 26 | 26 | 52
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 272 | 285 | 557
  Postmenopausal | 249 | 254 | 503
Hormone-receptor status [Count of Participants; unit: Participants]
  Positive | 349 | 344 | 693
  Negative | 170 | 192 | 362
  Unknown | 2 | 3 | 5
Surgery [Count of Participants; unit: Participants]
  Breast-conserving surgery: With radiation | 247 | 287 | 534
  Breast-conserving surgery: Without radiation | 24 | 24 | 48
  Mastectomy: With radiation | 20 | 22 | 42
  Mastectomy: Without radiation | 230 | 206 | 436

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) Events
Description: DFS is calculated from the date of randomization until the first date of recurrence local, regional or distant, second primary tumor or death.
Time Frame: 10 years
Measure: Number; unit: events
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 521 | 539
events | 127 | 112

2. Secondary Outcome: Overall Survival (OS)
Description: OS was determined from the date of randomization until the date of death for any reason.
  OS is calculated from the date of randomization up to the first date of death by any cause.
Time Frame: 10 years
Measure: Number; unit: Participants with mortality event
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 521 | 539
Participants with mortality event | 57 | 53

3. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Safety was assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 1.0.
Time Frame: Through study treatment, and average of 4 months
Population: The safety analysis was conducted on all patients who started at least one infusion of the study treatment (Arm A 519, and Arm B 532).
Measure: Number; unit: participants
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 519 | 532
participants
  Number patients with One AE | 519 | 532
  One G3-4 or severe treatment-emergent AE | 88 | 151
  One serious treatment-emergent AE | 22 | 119
  One serious G3-4 treatment-emergent AE | 10 | 55
  Number of patients discontinued due to AE | 4 | 25
  Number patients death due to AE | 0 | 1

4. Secondary Outcome: Best Score During Study for Global Health Status Scale
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) was used.
  Questionnaires were self-administered to patients during the 14 days prior to randomisation baseline, at six prospective time points corresponding to chemotherapy cycles, with the time window related to each chemotherapy cycle defined as the period between the day following the first chemotherapy dose of the corresponding cycle and the day of the first dose of the following cycle, and then at 44, 68 and 120 weeks of the study.
  The Global Health Status Scale has been used, which is calculated with questions 29 and 30 from the EORTC QLQ-C30. From this scale, the best score is the highest score observed during study (of all the questionnaires completed by patient). In this scale, scores range from 0 to 100 and a high score represents a high level of functioning or HRQoL.
Time Frame: 120 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 519 | 532
score on a scale | 79.30 (17.64) | 77.78 (18.87)

5. Secondary Outcome: Number of Disease Free Survival Events in Hormone-receptor Positive and Human Epidermal Growth Factor Receptor 2 (HER2) Positive Status Subgroup
Description: Hormone-receptor status and HER2 receptor status was analysed in Paraffin-embedded tumor samples obtained at the time of surgery, and were processed centrally. Disease-Free Survival (DFS) is defined as the interval from the date of randomization to the date of local, regional or metastatic relapse or the date of second primary cancer or death from any cause whichever occurs first.
Time Frame: 10 year
Measure: Number; unit: events
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 28 | 30
events | 6 | 6

6. Secondary Outcome: Disease Free Survival in Hormonal Receptor Positive and HER2 Negative Subgroup
Description: as for outcome 5
Time Frame: 10 year
Measure: Number; unit: events
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 209 | 220
events | 50 | 37

7. Secondary Outcome: Disease Free Survival in Hormonal Receptor Negative and HER2 Positive Subgroup
Description: Hormone-receptor status and HER2 receptor status was analysed in Paraffin-embedded tumor samples obtained at the time of surgery, and were processed centrally.
Time Frame: 10 year
Measure: Number; unit: events
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 24 | 22
events | 6 | 5

8. Secondary Outcome: Disease Free Survival in Hormonal Receptor Negative and HER2 Negative Subgroup
Description: as for outcome 5
Time Frame: 10 year
Measure: Number; unit: events
Arm/Group | Arm A: FAC | Arm B: TAC
Number analyzed (Participants) | 92 | 103
events | 29 | 28

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 10 years. Adverse Events were assessed for an average of 4 months
Description: The safety analysis were conducted on all patients who started at least one infusion of the study treatment.
Arm/Group | Arm A: FAC | Arm B: TAC
All-Cause Mortality (participants affected / at risk) | 57/519 | 53/532
Serious Adverse Events (participants affected / at risk) | 21/519 | 119/532
Other Adverse Events (participants affected / at risk) | 519/519 | 532/532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: FAC (N=519) | Arm B: TAC (N=532)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Blood bilirubin (Blood and lymphatic system disorders) | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 1
Breast infection (Reproductive system and breast disorders) | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Carotid artery thrombosis (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Erysipelas (Skin and subcutaneous tissue disorders) | 0 | 1
Ear infection (Ear and labyrinth disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Febrile neutropenia (Investigations) | 0 | 3
Fever in absence of infection (General disorders) | 12 | 68
General physical health deterioration (General disorders) | 0 | 1
Hypersensitivity (Nervous system disorders) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Oedema peripheral (Vascular disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Pancreatitis (Metabolism and nutrition disorders) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Thrombosis (Vascular disorders) | 0 | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: FAC (N=519) | Arm B: TAC (N=532)
Alopecia (Skin and subcutaneous tissue disorders) | 508 | 514
Asthenia (General disorders) | 305 | 387
Nausea (Gastrointestinal disorders) | 387 | 379
Stomatitis (Gastrointestinal disorders) | 265 | 292
Vomiting (Gastrointestinal disorders) | 294 | 292
Diarrhoea (Gastrointestinal disorders) | 70 | 147
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 123
Amenorrhoea (Reproductive system and breast disorders) | 70 | 121
Pain (General disorders) | 80 | 118
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 108
Conjunctivitis (Eye disorders) | 104 | 108
Menstruation irregular (Reproductive system and breast disorders) | 90 | 103
Nail disorder (Skin and subcutaneous tissue disorders) | 77 | 102
Oedema peripheral (Vascular disorders) | 19 | 101
Skin disorder (Skin and subcutaneous tissue disorders) | 51 | 96
Pyrexia (General disorders) | 46 | 90
Abdominal pain upper (Gastrointestinal disorders) | 71 | 88
Decreased appetite (General disorders) | 69 | 88
Dysgeusia (Nervous system disorders) | 71 | 85
Peripheral Sensory Neuropathy (Nervous system disorders) | 38 | 83
Hot flush (Reproductive system and breast disorders) | 54 | 74
Dyspepsia (Gastrointestinal disorders) | 50 | 57
Neutropenia (Blood and lymphatic system disorders) | 9 | 33
Weight increased (General disorders) | 10 | 29
Insomnia (Psychiatric disorders) | 24 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 26
Affective disorder (Psychiatric disorders) | 28 | 25
Lacrimation increased (Eye disorders) | 18 | 24
Bone pain (General disorders) | 1 | 18
Peripheral motor neuropathy (Nervous system disorders) | 2 | 18
Back pain (General disorders) | 6 | 17
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Lymphoedema (Vascular disorders) | 3 | 13
Arrhythmia (Cardiac disorders) | 6 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Haemorrhoids (Gastrointestinal disorders) | 6 | 11
Urinary tract infection (Infections and infestations) | 10 | 11
Erythema (Skin and subcutaneous tissue disorders) | 5 | 10
Chest pain (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Flatulence (Gastrointestinal disorders) | 2 | 6
Photophobia (Nervous system disorders) | 1 | 6
Vaginal infection (Infections and infestations) | 1 | 5
Fatigue (General disorders) | 7 | 4
Metrorrhagia (Reproductive system and breast disorders) | 2 | 4
Hyperhidrosis (General disorders) | 1 | 3
Infection (Infections and infestations) | 0 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 3
Visual impairment (Nervous system disorders) | 1 | 3
Herpes zoster (Infections and infestations) | 3 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Anal abscess (Gastrointestinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less